CLINICAL TRIAL: NCT04519281
Title: Role of Preoperative IV Administration of Vitamin C in Patients at Risk for Cardiac Vasoplegia After Cardiopulmonary Bypass
Brief Title: Role of Vitamin C in Cardiac Vasoplegia After Cardiopulmonary Bypass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham Mostafa Ahmed Alkady, Prof. A. Dr., Cairo University
Other Study IDs: N-17-2020
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: to Study the Effect of Vitamin C Administration on the Amount and the Time of Weaning of Noradrenaline Given Post-operatively to Patients After CPB
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group (A): consists of 50 patients undergoing open heart surgeries who will receive IV ascorbic acid
  Interventions: Drug: IV of vitamin C
- Group (B): consists of 50 patients undergoing open heart surgeries who will not receive ascorbic acid or will receive a placebo (Control Group).

INTERVENTIONS:
Drug: IV of vitamin C — administration of high-dose of IV vitamin C perioperatively
  Groups: Group (A)

SUMMARY:
This is a parallel group double-blind, randomized-controlled trial with 1:1 randomization ratio which will be conducted over a period of 6 months to study the effect of vitamin C administration on the amount of noradrenaline given post-operatively to patients after CPB. Two groups will be included; Group (A) patients undergoing open heart surgeries who will receive IV ascorbic acid (treatment group) and Group (B) patients undergoing open heart surgeries who will not receive ascorbic acid or will receive a placebo (control group). Each patient will be subjected to assessments of the doses of noradrenaline given from the end of surgery until weaning as well as hemodynamics in the first 2 hours and then at intervals of 6 hours up to 3 days following surgery.

DETAILED DESCRIPTION:
Background and Rationale:

Cardiac vasoplegia is a known phenomenon after cardiopulmonary bypass (CPB) occurring in up to 44% of patients. Severe forms of such condition refractory to vasopressors are associated with poor outcomes. New agents e.g. ascorbic acid that can alter the systemic vascular resistance in cardiac vasoplegia have been suggested as an attempt to avoid or at least reduce the use of IV vasopressors and their induced systemic hypo-perfusion.

Objectives :

* Primary objective: to study the effect of vitamin C administration on the amount of noradrenaline given post-operatively to patients after CPB
* Secondary objectives: to study the effect of vitamin C administration on the time to weaning from noradrenaline

Study population & Sample size :

Patients undergoing cardiac surgeries with CPB having risk factors for cardiac vasoplegia like diabetes mellitus and chronic renal failure.

50 patients will be needed in each group (treatment and control)

Study Design :

A parallel group double-blind, randomized-controlled trial, with 1:1 randomization ratio 2 groups will be included;

-Group (A) patients undergoing open heart surgeries who will receive IV ascorbic acid. -Group (B) patients undergoing open heart surgeries who will not receive ascorbic acid or will receive a placebo (Control Group).

Methods :

Each patient will be subjected to the following assessments:

-Pre-operative patient characteristics: demographic data, co-morbidities, pre-operative echo findings,… -Intra-operative details: procedures, time parameters,… the doses of noradrenaline given from the end of surgery until weaning or death and hemodynamics in the first 2 hours and then at intervals of 6 hours up to 3 days following surgery. -Postoperative data: echo parameters, patient outcome, time of discharge,…

Outcome parameter (s):

-Primary outcome: the area under the dose-time curve of noradrenaline -Secondary outcome measures: the duration of vasopressor (noradrenaline) infusion till weaning up to 3 days following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgeries with CPB having risk factors for cardiac vasoplegia like diabetes mellitus and chronic renal failure.

Exclusion Criteria:

* Patients who undergo surgeries without cardiopulmonary bypass (off-pump)
* Patients undergoing surgeries for congenital cardiac disease
* Patients performing heart transplantation and combined cardiac surgeries
* Patients with low pre-operative left ventricular ejection fraction (LVEF)
* Patients refusing to participate
* Patients who receive vasopressors other than noradrenaline

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A parallel group double-blind, randomized-controlled trial, with 1:1 randomization ratio 2 groups will be included;
  * Group (A) consists of 50 patients undergoing open heart surgeries who will receive IV ascorbic acid.
  * Group (B) consists of 50 patients undergoing open heart surgeries who will not receive ascorbic acid or will receive a placebo (Control Group).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
amount of noradrenaline need | 3 days
  to study the effect of vitamin C administration on the amount of noradrenaline given post-operatively to patients after CPB

SECONDARY OUTCOMES:
duration of noradrenaline need | 3 days
  to study the effect of vitamin C administration on the time to weaning from noradrenaline

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Clinical outcomes are to be shared

REFERENCES:
- [Background] Omar S, Zedan A, Nugent K. Cardiac vasoplegia syndrome: pathophysiology, risk factors and treatment. Am J Med Sci. 2015 Jan;349(1):80-8. doi: 10.1097/MAJ.0000000000000341. PMID 25247756
- [Background] Fischer GW, Levin MA. Vasoplegia during cardiac surgery: current concepts and management. Semin Thorac Cardiovasc Surg. 2010 Summer;22(2):140-4. doi: 10.1053/j.semtcvs.2010.09.007. PMID 21092891
- [Background] Wieruszewski PM, Nei SD, Maltais S, Schaff HV, Wittwer ED. Vitamin C for Vasoplegia After Cardiopulmonary Bypass: A Case Series. A A Pract. 2018 Aug 15;11(4):96-99. doi: 10.1213/XAA.0000000000000752. PMID 29634537